CLINICAL TRIAL: NCT03773198
Title: Effectiveness of Energy Resonance by Skin Stimulation in the Management of Anxious Patients Who Require Scheduled Orthopaedic Surgery
Acronym: ERESCAO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DAUVERGNE APPARA 2017
Record Dates: First submitted 2018-12-04; First posted 2018-12-12 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Patient Requiring Scheduled Conventional Orthopedic Surgical Intervention of the Upper or Lower Limb
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCS Group (Experimental)
  Interventions: Other: Energy Resonance through Cutaneous Stimulation; Other: questionnaires
- Control Group (Placebo Comparator)
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: Energy Resonance through Cutaneous Stimulation — The ERCS method involves "listening" to the body by applying fingers to the acupuncture skin points, developed according to the energy imbalance caused by illness, pain and emotional disorders.
  Arms: ERCS Group
Other: questionnaires — Measurement of anxiety-trait and state-anxiety (Spielberger), pain ( numerical scale) and satisfaction (numerical satisfaction scale)

SUMMARY:
The need for a surgical procedure may cause a patient to experience reactive anxiety. This reaction is appropriate if it is of low to moderate intensity. On the other hand, various studies have shown that postoperative awakening is more complicated if the patient experiences major preoperative anxiety. Thus, reducing anxiety could be a tool for preventing chronic pain.

For several years now, the investigator's facility has been implementing Energy Resonance through Cutaneous Stimulation (ERCS), a method based on "listening" to the body's vibrations through the fingers on points based on the mapping of meridians in Chinese medicine.

ERCS practitioners have noted the benefits of this method, particularly in soothing patients. It therefore seems necessary to detect and manage this anxiety beforehand and ERCS seems appropriate in this situation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given oral consent
* Adult patient requiring scheduled conventional orthopedic surgery of the upper limb (wrist, elbow, shoulder) or lower limb (ankle, foot, knee, hip)

Exclusion Criteria:

* Patient not affiliated to a national health insurance system,
* Patient subject to a legal protection measure (curatorship, guardianship)
* Patient subject to a justice protection measure
* Pregnant, parturient or breastfeeding woman
* Patient unable to give consent
* Minor
* Patient with a pace maker
* Patient with cognitive problems: Alzheimer's, senile dementia
* Patient who has already received ERCS as part of surgery
* Patient who does not speak or understand French
* Patient with psychiatric disorders: major depression, bipolar disorder, addictive disorders, psychotic disorders (psychosis, schizophrenia, acute delirium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
anxiety-state | During the surgical procedure
  Evolution of the patient's anxiety, between the entry and exit of the surgical department measured by the Spielberger state anxiety inventory, which is intended to evaluate an emotional reaction at a given time represented here by the operating room.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France